CLINICAL TRIAL: NCT06561984
Title: Effect of Antenatal Education on Pregnant Women's Knowledge, Attitude and Preferences of Delivery Mode
Brief Title: Effect of Antenatal Education on Knowledge,Attitude and Preferences Taward Delivery Modes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Hassan Ragab Elshrqawy, Assistant lecturer, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Antenatal Education
Record Dates: First submitted 2024-08-11; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Antenatal Education; Modes of Delivery
Keywords: Antenatal Education, Knowledge, attitude, Mode of delivery
MeSH Terms: conditions — Behavior | interventions — Prenatal Education

STUDY DESIGN:
Intervention Model Description: The intervention group will receive educational sessions regarding modes of delivery, while the control group will receive the routine antenatal care only in the antenatal clinics
Who Masked: Participant
Masking Description: The intervention group will receive educational sessions regarding modes of delivery, while the control group will receive the routine antenatal care only in the antenatal clinics
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive antenatal educational sessions regarding modes of delivery in addition to the routine care in the antenatal clinic
  Interventions: Behavioral: antenatal education
- Control group (No Intervention): The control group will receive only the routine care in the antenatal clinic

INTERVENTIONS:
Behavioral: antenatal education — Giving educational sessions to the intervention group regarding modes of delivery
  Arms: Intervention group

SUMMARY:
The aim of the current study is to assess the effect of antenatal education on pregnant women's knowledge, attitude, and preferences of delivery mode.

DETAILED DESCRIPTION:
This study employed a quasi-experimental design with intervention and control group. The purposive sample will consisted of 140 pregnant women who attended for prenatal care for follow up at the previously mentioned setting. The main objective of the study will to examine the effect of antenatal education on pregnant women's knowledge, attitude, and preferences toward the mode of delivery.

In order to accomplish the study's aim, the following research hypothesis is developed:

Hypothesis 1. Pregnant women who receive antenatal education will have a higher level of knowledge and positive attitude regarding the mode of delivery than those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are 18 to 35 years old.
* A singleton pregnancy in the third
* Primigravida and pregnant women with a history of one prior elective cesarean section at least two years between pregnancies.

Exclusion Criteria:

* Pregnant women who has any indication of a cesarean section or obstetrical issues that have arisen during the present pregnancy
* Pregnant woman who suffer from psychological illness.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Structured Interviewing Questionnaire. | 6 months
  This tool was designed by the researcher after an extensive review of the related national and international literature and was filled by the researcher It consists of three parts:
  Part I: Studied pregnant women's general characteristics including age, educational level of the mother and husband, residence, etc…).
  Part II: Obstetrical history of the studied pregnant women including gravidity, parity, history of abortion, type of previous C.S, inter-pregnancy interval, etc…).
  Part III: Knowledge of the studied pregnant women toward mode of delivery.
Tool II: Attitude of the studied pregnant women toward mode of delivery questionnaire | 6 months
  It was developed by the researcher. Its primary objective was to assess pregnant women attitude toward delivery mode, it consists of two parts:
  Part I: Attitude of the studied pregnant women toward vaginal delivery:
  Part II: Attitude of the studied pregnant women toward Cesarean section:
Tool III: Studied pregnant women's preference of delivery mode sheet. | 6 months
  The researcher developed this tool after reviewing the relevant literature (Elgzar, Alshahrani, & Ibrahim, 2023) to assess pregnant women preference of delivery mode. It included two items (the type of delivery mode as normal vaginal delivery or cesarean section and causes for choosing this mode of delivery, including labor pain, the cost, doctor preference, health beliefs regarding mode of delivery, the most common mode of delivery, having previous knowledge toward the mode of delivery, and having knowledge from an educational program, etc…).

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elshrqawy, Assist. lec, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Background] Akinlusi FM, Olayiwola AA, Rabiu KA, Oshodi YA, Ottun TA, Shittu KA. Prior childbirth experience and attitude towards subsequent vaginal birth after one caesarean delivery in Lagos, Nigeria: a cross-sectional study. BMC Pregnancy Childbirth. 2023 Jan 30;23(1):82. doi: 10.1186/s12884-023-05348-4. PMID 36717780
- [Background] AlSomali Z, Bajamal E, Esheaba O. The Effect of Structured Antenatal Education on Childbirth Self-Efficacy. Cureus. 2023 May 21;15(5):e39285. doi: 10.7759/cureus.39285. eCollection 2023 May. PMID 37223341
- [Background] Grobman WA, Sandoval GJ, Rice MM, Chauhan SP, Clifton RG, Costantine MM, Gibson KS, Metz TD, Parry S, Reddy UM, Rouse DJ, Saade GR, Simhan HN, Thorp JM Jr, Tita ATN, Yee L, Longo M, Landon MB; of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prediction of vaginal birth after cesarean using information at admission for delivery: a calculator without race or ethnicity. Am J Obstet Gynecol. 2024 Mar;230(3S):S804-S806. doi: 10.1016/j.ajog.2023.02.008. Epub 2023 Jul 14. No abstract available. PMID 38180754
- [Background] Gebremichael MA, Lema TB. Prevalence and Predictors of Knowledge and Attitude on Optimal Nutrition and Health Among Pregnant Women in Their First Trimester of Pregnancy. Int J Womens Health. 2023 Sep 4;15:1383-1395. doi: 10.2147/IJWH.S415615. eCollection 2023. PMID 37692922
- [Background] Al-Rifai RH, Elbarazi I, Ali N, Loney T, Oulhaj A, Ahmed LA. Knowledge and Preference Towards Mode of Delivery among Pregnant Women in the United Arab Emirates: The Mutaba'ah Study. Int J Environ Res Public Health. 2020 Dec 23;18(1):36. doi: 10.3390/ijerph18010036. PMID 33374611
- [Background] Zewude B, Siraw G, Adem Y. The Preferences of Modes of Child Delivery and Associated Factors Among Pregnant Women in Southern Ethiopia. Pragmat Obs Res. 2022 Jul 15;13:59-73. doi: 10.2147/POR.S370513. eCollection 2022. PMID 35873720
- [Background] Elgzar WT, Alshahrani MS, Ibrahim HA. Mode of delivery preferences: the role of childbirth fear among nulliparous women. Front Psychol. 2023 Nov 16;14:1221133. doi: 10.3389/fpsyg.2023.1221133. eCollection 2023. PMID 38034315
- [Derived] El-Shrqawy EH, Elnemer A, Mohamed Elsayed H. Effect of antenatal education on pregnant women;s knowledge, attitude and preferences of delivery mode. BMC Pregnancy Childbirth. 2024 Nov 12;24(1):740. doi: 10.1186/s12884-024-06922-0. PMID 39533248